CLINICAL TRIAL: NCT01396148
Title: A PHASE I/II STUDY OF SUNITINIB IN YOUNG PATIENTS WITH ADVANCED GASTROINTESTINAL STROMAL TUMOR
Brief Title: A Study of Sunitinib In Young Patients With Advanced Gastrointestinal Stromal Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A6181196; 2011-002008-33 (EudraCT Number)
Record Dates: First submitted 2011-07-13; First posted 2011-07-18 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Children and young adults with GIST; sunitinib malate; pharmacokinetics; tumor response; overall survival; tumor KIT mutation status
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Children with GIST (Experimental): children ages 6yrs-<18yrs
  Interventions: Drug: sunitinib malate dose escalation
- Young adults with GIST (Experimental): young adults ages 18yrs-<21 yrs
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate dose escalation — sunitinib starting dose will be 15mg/m^2 daily on a 4 weeks on/2 weeks off schedule (Schedule 4/2).
  Arms: Children with GIST
Drug: sunitinib malate — sunitinib 50mg daily on Schedule 4/2
  Arms: Young adults with GIST

SUMMARY:
Children and young adults with gastrointestinal stromal tumors (GIST) will be treated with sunitinib. The safety (including pharmacokinetics) and tolerability of sunitinib will be studied in these patients. In addition, tumor responses and overall survival will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of GIST.
* Patients must have demonstrated either disease progression or intolerance to imatinib mesylate, have non-mutant Stem Cell Factor Receptor gene (KIT) GIST, or cannot obtain imatinib in their country
* Measurable by Response Evaluation Criterion in Solid Tumors (RECIST) or evaluable disease.

Exclusion Criteria:

* Current treatment with another investigational agent.
* Prior sunitinib treatment.
* Prior therapy with known risk for cardiovascular complications.

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (3):
  - Children's Center for Cancer and Blood Diseases, Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Boston, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - FN Brno, Brno
  - Masarykuv onkologicky ustav, Brno
- France (3):
  - CHU de La Timone, Hopital enfants, Marseille
  - Hopital d'Enfants de la Timone, Marseille
  - Hopital de la Timone, Marseille

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Wang E, DuBois SG, Wetmore C, Verschuur AC, Khosravan R. Population Pharmacokinetics of Sunitinib and its Active Metabolite SU012662 in Pediatric Patients with Gastrointestinal Stromal Tumors or Other Solid Tumors. Eur J Drug Metab Pharmacokinet. 2021 May;46(3):343-352. doi: 10.1007/s13318-021-00671-7. Epub 2021 Apr 14. PMID 33852135
- [Derived] Verschuur AC, Bajciova V, Mascarenhas L, Khosravan R, Lin X, Ingrosso A, Janeway KA. Sunitinib in pediatric patients with advanced gastrointestinal stromal tumor: results from a phase I/II trial. Cancer Chemother Pharmacol. 2019 Jul;84(1):41-50. doi: 10.1007/s00280-019-03814-5. Epub 2019 Apr 20. PMID 31006038
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181196&StudyName=A%20Study%20of%20Sunitinib%20In%20Young%20Patients%20With%20Advanced%20Gastrointestinal%20Stromal%20Tumor

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib: Participants received Sunitinib capsules orally at a dose based on body surface area (BSA) (minimum dose of 15 milligram/ meter square [mg/m^2] up to a maximum dose of 30 mg/m^2) once daily, from Day 1 to 28 in each treatment cycle of 42 days (up to a maximum of 18 cycles) until completion of study treatment, disease progression, unacceptable toxicity, required a treatment rest (greater than [>4] weeks), withdrawal of participant consent, or if other withdrawal criteria were met.
Period: Overall Study
Arm/Group | Sunitinib
Started | 6
Completed | 5
Not Completed | 1
Not completed — Patient Decision | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all enrolled participants regardless of what treatment, if any, was received.
Arm/Group | Sunitinib
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 5
  Asian | 1

OUTCOME MEASURES:

1. Primary Outcome: Estimated Steady-State Maximum Plasma Concentration (Cmax,ss) of Sunitinib and Its Metabolite
Description: Estimated steady-state maximum plasma concentration (Cmax,ss) of Sunitinib and its metabolite SU012662. Summarized data for all time points was reported.
Time Frame: pre-dose on Day 1, Day 12-18 and Day 25-29 of Cycle 1,2, 3 and 2, 4, 6, 8 hours post-dose on Day 1 Cycle 1
Population: The PK population included all treated participants with at least one PK observation.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Sunitinib
Number analyzed (Participants) | 6
nanograms per milliliter (ng/mL)
  Sunitinib | 37.98 (12.91)
  SU012662 | 14.55 (3.04)

2. Primary Outcome: Estimated Area Under the Plasma Concentration Versus Time Curve From Time Zero to 24 Hours Post Dose AUC(0-24) of Sunitinib and Its Metabolite
Description: Estimated area under the plasma concentration versus time curve from time zero to 24 hours post dose (AUC24) of Sunitinib and its metabolite SU012662. Summarized data for all time points was reported.
Time Frame: pre-dose on Day 1, Day 12-18 and Day 25-29 of Cycle 1,2, 3 and 2, 4, 6, 8 hours post-dose on Day 1 Cycle 1
Population: The PK population included all treated participants with at least one PK observation.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr)/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 6
nanogram*hour per milliliter (ng*hr)/mL
  Sunitinib | 812.59 (273.37)
  SU012662 | 336.78 (74.15)

3. Primary Outcome: Estimated Oral Clearance (CL/F) of Sunitinib and Its Metabolite
Description: SU012662 is the metabolite of Sunitinib. Oral clearance (CL/F) is a quantitative measure of the rate at which a drug substance is removed from the blood (CL) normalized by the oral bioavailability of the drug (F). Summarized data for all time points was reported.
Time Frame: pre-dose on Day 1, Day 12-18 and Day 25-29 of Cycle 1,2, 3 and 2, 4, 6, 8 hours post-dose on Day 1 Cycle 1
Population: The PK population included all treated participants with at least one PK observation.
Measure: Mean (Standard Deviation); unit: Liters per hour (L/hr)
Arm/Group | Sunitinib
Number analyzed (Participants) | 6
Liters per hour (L/hr)
  Sunitinib | 26.37 (7.62)
  SU012662 | 12.85 (3.11)

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Sunitinib and Its Metabolite
Description: SU012662 is the metabolite of Sunitinib.
Time Frame: Cycle 1 Day 1: pre-dose, 2, 4, 6, and 8 hours post-dose
Population: The PK population included all treated participants with at least one PK observation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Sunitinib
Number analyzed (Participants) | 6
nanograms per milliliter (ng/mL)
  Sunitinib | 17.58 (32)
  SU012662 | 2.342 (18)

5. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Sunitinib and Its Metabolite
Description: SU012662 is the metabolite of Sunitinib.
Time Frame: Cycle 1 Day 1: pre-dose, 2, 4, 6, and 8 hours post-dose
Population: The PK population included all treated participants with at least one PK observation.
Measure: Median (Full Range); unit: hours
Arm/Group | Sunitinib
Number analyzed (Participants) | 6
hours
  Sunitinib | 8 [4 to 8]
  SU012662 | 8 [4 to 8]

6. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 8 Hours Post Dose AUC(0-8) for Sunitinib and Its Metabolite
Description: AUC(0-8) was defined as area under the plasma concentration time-curve from time zero to 8 hours post dose. SU012662 is the metabolite of Sunitinib.
Time Frame: Cycle 1 Day 1: pre-dose, 2, 4, 6, and 8 hours post-dose
Population: The PK population included all treated participants with at least one PK observation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*hr)/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 6
nanograms*hour per milliliter (ng*hr)/mL
  Sunitinib | 77.49 (42)
  SU012662 | 10.11 (37)

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to end of study (up to Cycle 18) that were absent before treatment or that worsened relative to pretreatment state. AEs included both non-serious adverse events (AEs) and SAEs.
Time Frame: Baseline up to end of study (up to Cycle 18, each cycle was of 42 days)
Population: The as-treated population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 6
participants
  AEs | 6
  SAEs | 0

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) Greater Than or Equal to (>=) Grade 3, Based on National Cancer Institute (NCI) Common Terminology Criteria (CTC) for AEs (CTCAE), Version 4.0
Description: An AE is any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. As per NCI CTCAE, Grade 3 events =medically significant but not immediately life-threatening, unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment, Grade 4 events =participant to be in imminent danger of death. Grade 5 events =death. Treatment-emergent events are events between first dose of study drug and up to end of study (up to Cycle 18) that were absent before treatment or that worsened relative to pretreatment state. Number of participants with AEs of any of the Grade 3 or above (Grade 4, 5) were reported.
Time Frame: Baseline up to end of study (up to Cycle 18, each cycle was of 42 days)
Population: The as-treated population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 6
participants | 5

9. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both non-serious adverse events (AEs) and SAEs.
Time Frame: Baseline up to end of study (up to Cycle 18, each cycle was of 42 days)
Population: The as-treated population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 6
participants
  AEs | 6
  SAEs | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Criteria for clinically significant laboratory abnormalities: Hemoglobin (Hb), hematocrit: less than (<) 0.8*lower limit of normal (LLN), platelet: <75 or greater than (>) 700*10^3/millimeter (mm)^3*upper limit of normal (ULN), leukocyte: <2.5 or >17.5*10^3/mm^3*ULN; total bilirubin 1.5*ULN, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gamma-glutamyl transferase: >3.0*ULN, total protein, albumin: <0.8*LLN or >1.2*ULN ;blood urea nitrogen, creatinine: >1.3*ULN, uric acid >1.2*ULN; sodium <0.95*LLN or >1.05*ULN, potassium, calcium: <0.9*LLN or >1.1*ULN, albumin, total protein <0.8*LLN or >1.2*ULN; glucose <0.6*LLN or >1.5*ULN, creatine kinase >2.0*ULN; urine (red blood cell, white blood cell >6/high power field).
Time Frame: Baseline up to end of study (up to Cycle 18, each cycle was of 42 days)
Population: The as-treated population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 6
participants | 0

11. Secondary Outcome: Number of Participants With Objective Response
Description: Objective response in participants was defined as the number of participants with confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Confirmed response were those that persisted on repeat imaging study for at least 4 weeks after initial documentation of response. CR was defined as disappearance of all lesions (target and non-target). PR was defined as at least 30 percentage (%) decrease in the sum of the longest dimensions of target lesions taking as a reference the baseline sum longest dimensions, with non-target lesions not increased or absent.
Time Frame: Baseline until disease progression or discontinuation from the study, or death, whichever occurred first (maximum duration: up to Cycle 18; each cycle was of 42 days)
Population: The full analysis set included all enrolled participants regardless of what treatment, if any, was received.
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 6
participants
  Complete response | 0
  Partial response | 0

12. Secondary Outcome: Duration of Response
Description: Duration of response was defined as time (in months) from the first documentation of objective tumor response (confirmed CR or PR) to the first documentation of disease progression or death due to any cause. Confirmed response were those that persisted on repeat imaging study for at least 4 weeks after initial documentation of response. CR was defined as disappearance of all lesions (target and non-target). PR was defined as at least 30% decrease in the sum of the longest dimensions of target lesions taking as a reference the baseline sum longest dimensions, with non-target lesions not increased or absent. Progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: as for outcome 11
Population: Analysis was performed on a subset of FAS which included participants who had a confirmed CR or PR. Since, none of the participants had confirmed CR or PR, hence duration of response was not analyzed.
Arm/Group | Sunitinib
Number analyzed (Participants) | 0

13. Secondary Outcome: Progression-Free Survival
Description: Progression free survival was defined as time (in months) from date of enrollment to the first documentation of disease progression or to death (due to any cause), whichever occurred first. Progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: as for outcome 11
Population: The full analysis set included all enrolled participants regardless of what treatment, if any, was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib
Number analyzed (Participants) | 6
months | 5.8 [2.3 to NA] — The upper limit of the 95% CI was not estimable due to the small number of events.

14. Secondary Outcome: Overall Survival
Description: Overall survival was defined as time (in months) from enrollment to the date of death due to any cause. Analysis was performed using Kaplan-Meier method.
Time Frame: Baseline until death or discontinuation from the study whichever occurred first (maximum duration: up to Cycle 18; each cycle was of 42 days)
Population: The full analysis set included all enrolled participants regardless of what treatment, if any, was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib
Number analyzed (Participants) | 6
months | NA [NA to NA] — There were no deaths in study population, hence OS was not summarized using the Kaplan-Meier method.

15. Secondary Outcome: Number of Participants With Adverse Events Based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) for Pharmacokinetic (PK) Subgroups
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per NCI CTCAE version 4.0, Grade1= asymptomatic or mild symptoms, Grade 2= Moderate;local or noninvasive intervention indicated; Grade 3 events =medically significant but not immediately life-threatening, unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment, Grade 4 events =participant to be in imminent danger of death. Grade 5 events =death. Participants with any of the Grade 1 to Grade 5 AEs were reported. The PK evaluable participants were divided into 2 PK subgroups on Day 28 of Cycle 1: those with total drug (sunitinib + SU012662) trough plasma concentration (Ctrough) value less than (<) the median Ctrough value(lower exposure) and those with total drug (sunitinib + SU012662) Ctrough values greater than or equal to (>=) the median Ctrough value(higher exposure).
Time Frame: Cycle 1 Day 28 up to Cycle 3 (each cycle 42 days)
Population: The PK subgroup analysis set included all treated participants with at least 1 PK observation.
Measure: Number; unit: participants
Groups:
- Sunitinib: Lower Exposure: Participants who received Sunitinib capsules orally at a dose based on BSA (minimum dose of 15 mg/m^2 up to a maximum dose of 30 mg/m^2 once daily, from Day 1 to 28 in each treatment cycle of 42 days (up to a maximum of 18 cycles) and had total drug (sunitinib + SU012662) trough plasma concentration (Ctrough) < the median Ctrough value
- Sunitinib: Higher Exposure: Participants who received Sunitinib capsules orally at a dose based on BSA (minimum dose of 15 mg/m^2 up to a maximum dose of 30 mg/m^2 once daily, from Day 1 to 28 in each treatment cycle of 42 days (up to a maximum of 18 cycles) and had total drug (sunitinib + SU012662) trough plasma concentration (Ctrough) >= the median Ctrough value
Arm/Group | Sunitinib: Lower Exposure | Sunitinib: Higher Exposure
Number analyzed (Participants) | 3 | 3
participants
  Nausea | 0 | 2
  Vomiting | 0 | 1
  Diarrhoea | 0 | 2
  Fatigue | 0 | 1
  Palmar-Plantar Erythrodysaesthesia Syndrome | 1 | 0
  Neutropenia | 2 | 1
  Thrombocytopenia | 1 | 1
  Lymphopenia | 0 | 0
  Hypertension | 0 | 0
  Anaemia | 1 | 0

16. Secondary Outcome: Pearson Correlation Coefficient Between Percent Change From Baseline in Laboratory Parameters With Total Drug (Sunitinib + SU012662) Concentration
Description: Pearson correlation coefficient between percent change from baseline in laboratory parameters with total drug (Sunitinib + SU012662) concentration were calculated on Day 28 of Cycles 1, 2, and 3. Laboratory parameters included absolute neutrophil count, platelet count, lymphocyte count and hemoglobin.
Time Frame: Baseline, Day 28 of Cycle 1, Cycle 2 and Cycle 3 (each cycle was of 42 days)
Population: The PK population included all treated participants with at least one PK observation.
Measure: Number; unit: correlation coefficient
Arm/Group | Sunitinib
Number analyzed (Participants) | 6
correlation coefficient
  Absolute Neutrophil Count: Cycle 1 Day 28 | -0.1870
  Absolute Neutrophil Count: Cycle 2 Day 28 | -0.5914
  Absolute Neutrophil Count: Cycle 3 Day 28 | -0.5536
  Platelet Count: Cycle 1 Day 28 | 0.0329
  Platelet Count: Cycle 2 Day 28 | -0.6424
  Platelet Count: Cycle 3 Day 28 | -0.6604
  Lymphocyte Count: Cycle 1 Day 28 | 0.1509
  Lymphocyte Count: Cycle 2 Day 28 | -0.4815
  Lymphocyte Count: Cycle 3 Day 28 | -0.2931
  Hemoglobin: Cycle 1 Day 28 | 0.9107
  Hemoglobin: Cycle 2 Day 28 | 0.4368
  Hemoglobin: Cycle 3 Day 28 | 0.2095

17. Secondary Outcome: Pearson Correlation Coefficient Between Percent Change From Baseline in Vital Sign Results With Total Drug (Sunitinib + SU012662) Concentration
Description: Pearson correlation coefficient between percent change from baseline in vital sign results with total drug (Sunitinib + SU012662) concentration were calculated on Day 28 of Cycles 1, 2, and 3. Vital signs included systolic blood pressure and diastolic blood pressure.
Time Frame: Baseline, Day 28 of Cycle 1, Cycle 2 and Cycle 3 (each cycle was of 42 days)
Population: The PK population included all treated participants with at least one PK observation.
Measure: Number; unit: correlation coefficient
Arm/Group | Sunitinib
Number analyzed (Participants) | 6
correlation coefficient
  Systolic Blood Pressure: Cycle 1 Day 28 | -0.3730
  Systolic Blood Pressure: Cycle 2 Day 28 | -0.8146
  Systolic Blood Pressure: Cycle 3 Day 28 | 0.2768
  Diastolic Blood Pressure: Cycle 1 Day 28 | 0.6854
  Diastolic Blood Pressure: Cycle 2 Day 28 | -0.3638
  Diastolic Blood Pressure: Cycle 3 Day 28 | 0.2634

18. Secondary Outcome: Number of Participants With Stable Disease (SD), Partial Response (PR), Complete Response (CR) and Progressive Disease (PD) for PK Sub-groups
Description: SD:when there is no sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PR: as at least 30% decrease in the sum of the longest dimensions of target lesions taking as a reference the baseline sum longest dimensions, with non-target lesions not increased or absent. CR: disappearance of all lesions (target and non-target). PD:at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). Participants with SD, PR, CR and PD responses were assessed according to 2 PK subgroups created on Day 28 of Cycle 1: those with total drug (sunitinib + SU012662) trough plasma concentration (Ctrough) value less than (<) the median Ctrough value(lower exposure) and those with total drug (sunitinib + SU012662) Ctrough values greater than or equal to (>=) the median Ctrough value(higher exposure).
Time Frame: Baseline until disease progression or discontinuation from the study, or death, whichever occurred first(maximum duration: up to Cycle 18; each cycle was of 42 days)
Population: The PK population included all treated participants with at least 1 PK observation.
Measure: Number; unit: participants
Arm/Group | Sunitinib: Lower Exposure | Sunitinib: Higher Exposure
Number analyzed (Participants) | 3 | 3
participants
  Stable Disease | 1 | 2
  Partial Response | 0 | 0
  Complete Response | 0 | 0
  Progressive Disease | 2 | 1

19. Secondary Outcome: Progression Free Survival for PK Subgroups
Description: Progression free survival was defined as time (in months) from date of enrollment to the first documentation of disease progression or to death (due to any cause), whichever occurred first. Progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The PK evaluable participants were assessed according to 2 PK subgroups created on Day 28 of Cycle 1: those with total drug (sunitinib + SU012662) trough plasma concentration (Ctrough) value less than (<) the median Ctrough value(lower exposure) and those with total drug (sunitinib + SU012662) Ctrough values greater than or equal to (>=) the median Ctrough value(higher exposure).
Time Frame: as for outcome 11
Population: The PK population included all treated participants with at least one PK observation.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib: Lower Exposure | Sunitinib: Higher Exposure
Number analyzed (Participants) | 3 | 3
months | 2.6 [2.4 to NA] — The upper limit of the 95% CI was not estimable due to the small number of events | 9.0 [2.3 to NA] — The upper limit of the 95% CI was not estimable due to the small number of events

20. Secondary Outcome: Pearson Correlation Coefficient Between Progression Free Survival With Total Drug (Sunitinib + SU012662) Concentration
Description: Pearson correlation coefficient between Progression Free Survival (PFS) with total drug (Sunitinib + SU012662) concentration at Day 28 of Cycle 1 was calculated. PFS was defined as time (in months) from date of enrolment to the first documentation of disease progression or to death (due to any cause), whichever occurred first. Progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: Baseline until disease progression or discontinuation from the study, or death, whichever occurred first (maximum duration: up to Cycle 18; each cycle was of 42 days
Population: The PK population included all treated participants with at least one PK observation.
Measure: Number; unit: correlation coefficient
Arm/Group | Sunitinib
Number analyzed (Participants) | 6
correlation coefficient | 0.5904

21. Secondary Outcome: Estimated Sunitinib Plasma Concentration at Which 50% of the Maximum Effect (EC50) for Each Selected Efficacy Parameter (e.g., Sum of Largest Diameters for Target Tumors) Was Observed
Time Frame: Cycle 1 Day 1: pre-dose, 2, 4, 6, and 8 hours post-dose
Population: Due to low number of enrolled participants (n=6), there was insufficient data to perform any type of pharmacokinetic/pharmacodynamic modeling to obtain EC50 values, hence data is not reported.
Arm/Group | Sunitinib
Number analyzed (Participants) | 0

22. Secondary Outcome: Estimated Sunitinib Plasma Concentration at Which 50% of the Maximum Effect (EC50) for Each Selected Safety Endpoint (e.g., Absolute Neutrophil Count) Was Observed
Time Frame: Cycle 1 Day 1: pre-dose, 2, 4, 6, and 8 hours post-dose
Population: as for outcome 21
Arm/Group | Sunitinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (up to Cycle 18, each cycle was of 42 days)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Sunitinib
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=6)
Anaemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Palpitations (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Impaired gastric emptying (Gastrointestinal disorders) | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1
Lip discolouration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Sensitivity of teeth (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Hepatic haematoma (Hepatobiliary disorders) | 1
Ear infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase (Investigations) | 1
Blood phosphorus increased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Eosinophil count decreased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 4
Migraine (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/48/NCT01396148/Prot_000.pdf
  • Statistical Analysis Plan (2011-07-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT01396148/SAP_001.pdf